CLINICAL TRIAL: NCT00193856
Title: A Randomised Trial Investigating the Effect on Biochemical (PSA) Control and Survival of Different Durations of Adjuvant Androgen Deprivation in Association With Definitive Radiation Treatment for Localised Carcinoma of the Prostate.
Brief Title: RADAR Trial - Randomised Androgen Deprivation and Radiotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Hunter Medical Research Institute (HMRI) (Unknown); Health Research Council, New Zealand (Other); Novartis Pharmaceuticals (Industry); Cancer Society of New Zealand (Unknown); University of Newcastle, Australia (Other); Calvary Mater Newcastle, Australia (Other); Maitland Cancer Appeal (Unknown); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TROG 03.04; ACTRN12607000097448 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen Deprivation; Hormone Therapy; RadiotherapyBisphosphonate; Prostate Specific Antigen (PSA)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Active Comparator): LH-RH analogue for 5 months prior to and during first month of radiation treatment (total 6 mths)
  Interventions: Drug: Leuprorelin Acetate; Radiation: Conventional external beam therapy
- B (Active Comparator): LH-RH analogue for 5 months prior to and during first month of radiation treatment (total 6 months) + bisphosphonate therapy.
  Interventions: Drug: Leuprorelin Acetate; Drug: Zoledronic Acid; Radiation: Conventional external beam therapy
- C (Experimental): LH-RH analogue as for arm A, but continued for further 12 months (total 18 months)
  Interventions: Drug: Leuprorelin Acetate; Radiation: Conventional external beam therapy
- D (Experimental): LH-RH analogue as for arm A, but continued for further 12 months (total 18 months) + bisphosphonate therapy.
  Interventions: Drug: Leuprorelin Acetate; Drug: Zoledronic Acid; Radiation: Conventional external beam therapy

INTERVENTIONS:
Drug: Leuprorelin Acetate — LH-RH analogue (LH-RHa) (Leuprorelin acetate 22.5 mg) will be delivered as a depot injection every 3 months. This will be administered as an intramuscular injection (IMI).
Drug: Zoledronic Acid — Zoledronic acid 4 mg will be delivered as an intravenous infusion over 15 minutes once every 3 months for 18 months, in patients randomised to bisphosphonate therapy.
  Arms: B; D
Radiation: Conventional external beam therapy — The prescribed dose will be 66 Gy in 33 fractions of 2 Gy to the ICRU 50 point utilising a minimum of three fields with >= 6 MV photons.

SUMMARY:
The principal objectives of the RADAR trial is to address the hypotheses; 1) that 18 months androgen deprivation in conjunction with radiotherapy is superior to 6 months androgen deprivation prior to and during radiotherapy; 2) that 18 months Bisphosphonate therapy will prevent bone loss caused by androgen deprivation therapy and further reduce relapse risk by impeding the development of bony metastases.

DETAILED DESCRIPTION:
Traditionally androgen deprivation (by orchidectomy, or more recently by medication) has been reserved for the palliative treatment of men with advanced, incurable prostate cancer. However, evidence from large scale trials is beginning to suggest that androgen deprivation (AD) may be helpful in preventing relapse in patients with more localised disease who are treated surgically or by radiotherapy. Of the 8000 patients per annum who are treated with curative intent, one half (4000) have cancers where 'adjuvant' AD may be prescribed according to interpretation of the registered indications. There are, however, enormous variations in prescribing practices which reflect uncertainty as to the appropriate indications. An important issue is osteopenia.

The increasing use of AD in men with earlier stages of cancer, whose life expectancies exceed 3 years, has exposed many unwanted metabolic sequelae of prolonged AD, the most important being osteopenia. In 1996, with the funding support of the NHMRC and the pharmaceutical industry, TROG therefore launched a large randomised three-arm trial. Two of the arms repeated the two arms of the US Radiation Therapy Oncology Group (RTOG) 86.01 trial which, at the time, was showing early indications of benefit for the addition of two months maximal androgen deprivation (MAD), using Goserelin (Zoladex) and Flutamide, before radiation therapy and one month during. Since work from Canada had indicated that continued AD for periods longer than three months produced additional shrinkage of the prostatic tumour, the TROG 96.01 trial incorporated a third arm: six months MAD prior to and during radiotherapy. The trial completed its recruitment target of 800 eligible patients in early 2000. Although in August 2001 the median follow up time was still very short, a preliminary analysis indicated that significant increases in time to biochemical relapse had been produced by AD. In fact, the benefits of AD were independent of stage, tumour grade and initial PSA value which were confirmed also to predict time to biochemical failure. The hazard of relapse reduced to 0.75 (0.55 - 0.97, 95% confidence intervals) with 3 months AD, and still further to 0.6 (0.45 - 0.82) with six months AD.

Subsequent international developments in this area of research encouraged the design of a 'follow on' trial. A European Organisation for Research and Treatment of Cancer (EORTC) trial reported that 3 years of adjuvant ('post hoc') AD (using Goserelin alone), administered after radiotherapy, reduced relapse and improved survival in patients with locally advanced prostate cancer. The US Radiation Therapy Oncology Group (RTOG) 85.31 trial indicated that indefinite Goserelin administration after radiotherapy reduced treatment failure rates at all sites when compared with radiotherapy alone. The RTOG 92.02 trial showed that 24 months of adjuvant Goserelin also reduced failure rates in patients treated with 4 months of MAD prior to and during radiotherapy. Subset analyses of the RTOG trials, suggested that patients who gain most from prolonged AD in terms of survival are those with high grade cancers.

It was therefore logical for TROG to propose a second trial with the intention of finding out whether an additional 12 months of AD administered after radiotherapy (aka 'intermediate term' AD [ITAD]) would reduce relapse and mortality in patients treated with six months of AD prior to and during radiotherapy (aka 'short term' AD [STAD]) as in the 'best' arm of its first (96.01) trial. The availability of the potent bisphosphonate, zoledronic acid, also made it possible to find out whether or not osteopenia induced in the two arms of the proposed second trial would be prevented by a second random assignment to 18 months' bisphosphonate therapy (BP).

This is a randomised phase III multicentre clinical trial.

After informed consent is given and eligibility is checked patients will be randomised to one of four trial arms:

1. 6 months of androgen blockade with an LH-RH analogue (5 months before start of radiotherapy) (STAD),
2. 18 months of androgen blockade with an LH-RH analogue (starting 5 months before start of radiotherapy) (ITAD),
3. 18 months of therapy with zoledronic acid 4 mg by intravenous infusion every 3 months for 18 months beginning concurrently with STAD
4. 18 months of therapy with zoledronic acid beginning concurrently with ITAD.

Stratification will be according to the following criteria:

T2 / T3, 4 Gleason score 2 - 6 / 7+ Presenting PSA <10 / 10 - 20 / >20 Treatment centre

Radiation Treatment will be delivered using a conventional technique, unless the treatment centre of the participating clinician demonstrates an ability to deliver the treatment using a CRT, IMRT, or HDRB technique verified by the trial TACT.

Drug Treatment:

LH-RH analogue (LH-RHa) (Leuprorelin acetate 22.5 mg) will be delivered as a depot injection every 3 months. This will be administered as an Intramuscular injection (IMI).

Zoledronic acid 4 mg will be delivered as an intravenous infusion over 15 minutes once every 3 months for 18 months, in patients randomised to this therapy. No placebo therapy will be given to patients randomised to 'no bisphosphonate therapy' treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of adenocarcinoma of the prostate in the three months prior to randomisation
* Gleason primary and secondary pattern reported. If the volume of tumour in biopsies is too small for the pathologist to allocate a secondary pattern, the primary pattern alone is sufficient.
* Primary tumour stage T2b - 4 (UICC 2002), or T2a providing biopsies demonstrate Gleason score 7 or more, and presenting PSA 10 or more
* PSA value obtained within one month of randomisation
* No evidence of lymphatic or haematogenous metastases, as determined by negative chest x-ray, CT scan of abdomen and pelvis, and bone scan in the 3 months prior to randomisation
* ECOG performance status 0 - 1
* No concurrent medical conditions likely to significantly reduce prospects of 5 year survival
* Patient accessible to follow up at intervals specified in protocol
* Written informed consent given (signed by both patient and investigator prior to randomisation)

Exclusion Criteria:

* Previous or concurrent malignancy within previous 5 years except for non-melanomatous skin cancer
* Prostatectomy
* Prior pelvic radiotherapy
* Prior hormone treatment for prostate cancer
* Inability to complete self administered QOL questionnaire
* Prior bisphosphonate therapy
* Serum creatinine > 2 x ULN
* Osteoporosis resulting in >30% loss in vertebral height in one or more thoraco-lumbar vertebrae
* Liver disease resulting in ALT or AST levels >3 x ULN
* Prolonged continuous glucocorticoid therapy > 10 mg/day of prednisone equivalent (>6 months)
* Current treatment with bisphosphonate
* Inability to attend for follow-up at the Investigator's clinic

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1071 (Actual)
Dates: Start 2003-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Prostate cancer-specific mortality. | Two main endpoint analyses are planned when 6.5 and 10 years have elapsed from randomisation of the last participant

SECONDARY OUTCOMES:
Cumulative incidence of PSA progression | Two main endpoint analyses are planned when 6.5 and 10 years have elapsed from randomisation of the last participant
Cumulative incidence of local, distant and bony progression and associated patterns of clinical progression | Two main endpoint analyses are planned when 6.5 and 10 years have elapsed from randomisation of the last participant
All-cause mortality | Two main endpoint analyses are planned when 6.5 and 10 years have elapsed from randomisation of the last participant
Changes in bone mineral density and osteopenic fracture | One endpoint analysis is planned when 4.5 years have elapsed from randomisation of the last participant
Quality of life assessment | One endpoint analysis is planned when 3 years have elapsed from randomisation of the last participant
Treatment related morbidity | One endpoint analysis is planned when 4 years have elapsed from randomisation of the last participant
Cumulative incidence of secondary therapeutic intervention | Two main endpoint analyses are planned when 6.5 and 10 years have elapsed from randomization of the last participant

CONTACTS AND LOCATIONS:
Overall Officials: Jim Denham, FRANZCR, Study Chair — University of Newcastle, Australia
Locations (24):
- Australia (18):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Lismore Hospital, Lismore, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Nepean Cancer Care Centre, Penrith, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Illawarra Cancer Care Centre, Wollongong, New South Wales
  - Royal Brisbane Hospital, Herston, Queensland
  - Mater QRI, South Brisbane, Queensland
  - John Flynn Private Hospital, Tugun, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Launceston General Hospital, Launceston, Tasmania
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Andrew Love Cancer Care Centre, Geelong Hospital, Geelong, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- New Zealand (6):
  - Auckland Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Palmerston North Hospital, Palmerston North
  - Wellington Hospital, Wellington

REFERENCES:
- [Result] Haworth A, Kearvell R, Greer PB, Hooton B, Denham JW, Lamb D, Duchesne G, Murray J, Joseph D. Assuring high quality treatment delivery in clinical trials - Results from the Trans-Tasman Radiation Oncology Group (TROG) study 03.04 "RADAR" set-up accuracy study. Radiother Oncol. 2009 Mar;90(3):299-306. doi: 10.1016/j.radonc.2008.10.011. Epub 2008 Nov 18. PMID 19017549
- [Derived] Denham JW, Joseph D, Lamb DS, Spry NA, Duchesne G, Matthews J, Atkinson C, Tai KH, Christie D, Kenny L, Turner S, Gogna NK, Diamond T, Delahunt B, Oldmeadow C, Attia J, Steigler A. Short-term androgen suppression and radiotherapy versus intermediate-term androgen suppression and radiotherapy, with or without zoledronic acid, in men with locally advanced prostate cancer (TROG 03.04 RADAR): 10-year results from a randomised, phase 3, factorial trial. Lancet Oncol. 2019 Feb;20(2):267-281. doi: 10.1016/S1470-2045(18)30757-5. Epub 2018 Dec 19. PMID 30579763
- [Derived] Moulton CR, House MJ, Lye V, Tang CI, Krawiec M, Joseph DJ, Denham JW, Ebert MA. Prostate external beam radiotherapy combined with high-dose-rate brachytherapy: dose-volume parameters from deformably-registered plans correlate with late gastrointestinal complications. Radiat Oncol. 2016 Oct 31;11(1):144. doi: 10.1186/s13014-016-0719-2. PMID 27799048
- [Derived] Denham JW, Steigler A, Joseph D, Lamb DS, Spry NA, Duchesne G, Atkinson C, Matthews J, Turner S, Kenny L, Tai KH, Gogna NK, Gill S, Tan H, Kearvell R, Murray J, Ebert M, Haworth A, Kennedy A, Delahunt B, Oldmeadow C, Holliday EG, Attia J. Radiation dose escalation or longer androgen suppression for locally advanced prostate cancer? Data from the TROG 03.04 RADAR trial. Radiother Oncol. 2015 Jun;115(3):301-7. doi: 10.1016/j.radonc.2015.05.016. Epub 2015 Jun 10. PMID 26072289
- [Derived] Denham JW, Joseph D, Lamb DS, Spry NA, Duchesne G, Matthews J, Atkinson C, Tai KH, Christie D, Kenny L, Turner S, Gogna NK, Diamond T, Delahunt B, Oldmeadow C, Attia J, Steigler A. Short-term androgen suppression and radiotherapy versus intermediate-term androgen suppression and radiotherapy, with or without zoledronic acid, in men with locally advanced prostate cancer (TROG 03.04 RADAR): an open-label, randomised, phase 3 factorial trial. Lancet Oncol. 2014 Sep;15(10):1076-89. doi: 10.1016/S1470-2045(14)70328-6. Epub 2014 Aug 14. PMID 25130995
- [Derived] Denham JW, Wilcox C, Joseph D, Spry NA, Lamb DS, Tai KH, Matthews J, Atkinson C, Turner S, Christie D, Gogna NK, Kenny L, Duchesne G, Delahunt B, McElduff P. Quality of life in men with locally advanced prostate cancer treated with leuprorelin and radiotherapy with or without zoledronic acid (TROG 03.04 RADAR): secondary endpoints from a randomised phase 3 factorial trial. Lancet Oncol. 2012 Dec;13(12):1260-70. doi: 10.1016/S1470-2045(12)70423-0. Epub 2012 Nov 12. PMID 23151431
- [Derived] Denham JW, Wilcox C, Lamb DS, Spry NA, Duchesne G, Atkinson C, Matthews J, Turner S, Kenny L, Tai KH, Gogna NK, Ebert M, Delahunt B, McElduff P, Joseph D. Rectal and urinary dysfunction in the TROG 03.04 RADAR trial for locally advanced prostate cancer. Radiother Oncol. 2012 Nov;105(2):184-92. doi: 10.1016/j.radonc.2012.09.018. Epub 2012 Nov 3. PMID 23127770
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au